CLINICAL TRIAL: NCT03191916
Title: Transcranial Direct Current Stimulation (tDCS) to Improve Cognitive Function and Cognitive Fatigue in Parkinson's Patients
Brief Title: Transcranial Direct Current Stimulation for Cognitive Improvement in Parkinson's Patients
Acronym: tDCS
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sanford Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SH tDCS Parkinsons
Record Dates: First submitted 2017-04-28; First posted 2017-06-19 (Actual); Last update posted 2025-03-04 (Actual); Status verified 2025-02

CONDITIONS: Parkinson Disease
Keywords: Parkinson's Disease; tDCS; Cognitive function
MeSH Terms: conditions — Parkinson Disease | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned to an experimental group (receives stimulation) or a sham group (is set up with tDCS, but no stimulation is received)
Who Masked: Participant, Care Provider
Masking Description: The participant and their care provider will be blinded as to which intervention is being used.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- Experimental group (Experimental): The experimental group will receive 2 milliamps of anodal transcranial direct current stimulation for 20 minutes daily for 5 days.
  Interventions: Device: transcranial direct current stimulation
- Sham group (Sham Comparator): The sham group will be connected to the anodal transcranial direct current stimulation device daily for 5 days. During the 20 minute sessions, the participant will only receive stimulation for a 30-second ramp up period, at which point the stimulation will be discontinued for the remainder of the time.
  Interventions: Device: Sham (for transcranial direct current stimulation)

INTERVENTIONS:
Device: transcranial direct current stimulation — 2milliamps will be administered for 5 consecutive days for a duration of 20 minutes with electrode placement at the left dorsolateral prefrontal cortex.
  Other Names: Magstim; HDCstim; HDCkit
  Arms: Experimental group
Device: Sham (for transcranial direct current stimulation) — For 30 seconds the patient will experience a ramp up of the stimulation, after which point no stimulation will be transmitted for the remainder of the session. This will be administered for 5 consecutive days for a duration of 20 minutes with electrode placement at the left dorsolateral prefrontal cortex.
  Arms: Sham group

SUMMARY:
The investigators hypothesize that multi-session anodal tDCS (atDCS) of the left dorsolateral prefrontal cortex (LDLPFC) will induce long-lasting effects in improving cognitive function and reducing cognitive fatigue and fatigability in PD patients.

DETAILED DESCRIPTION:
Parkinson's disease (PD) is the second most common neurodegenerative disease (after Alzheimer's disease) and affects approximately one million people in the United States. Mild Cognitive Impairment (MCI) is very common even in early stages of PD. In addition to cognitive impairment, patients with PD also suffer cognitive fatigue (defined as the general sensation of difficulty in initiating cognitive activity) and cognitive fatigability (defined as "deterioration in the performance of attention tasks over an extended period of time"). Cognitive impairment, cognitive fatigue, and cognitive fatigability affect quality of life in patient with Parkinson's disease.

Transcranial direct current stimulation (tDCS) is a noninvasive and safe brain stimulation technique that has been shown to be effective in improving cognitive function in subjects with Parkinson's disease. During tDCS, low-voltage, low amplitude current is passed through a pair of surface electrodes placed over the areas of brain of interest.

The specific aim of this study is to examine if atDCS to LDLPFC at 2 milliamps (mA) for 20 minutes daily for 5 days will improve cognitive function and reduce cognitive fatigue and fatigability in PD patients with MCI. The study will examine if the effects may last for two weeks.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of PD with at least two of the four diagnostic criteria for PD (tremor, rigidity, bradykinesia, and postural instability)
* Meets criteria for MCI (21 ≤ MOCA scores ≤ 26)
* Must be able to consent

Exclusion Criteria:

* Patients with dementia (MOCA < 21)
* PD treatment using deep brain stimulation (DBS)
* Diagnosis of psychosis
* Diagnosis of multiple sclerosis
* Diagnosis of stroke
* Diagnosis of epilepsy
* Diagnosis of chronic obstructive pulmonary disease
* Diagnosis of congestive heart failure
* Diagnosis of renal failure
* Participants not fluent in English

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2015-10-19 (Actual); Primary Completion 2025-08-07 (Estimated); Study Completion 2025-08-31 (Estimated)

PRIMARY OUTCOMES:
Change in Reaction Time (RT) on contextual cueing computer task | 90 minutes; pre-test during the second research visit, post-test on 6th research visit after 5 consecutive days of tDCS, a follow up test on the 7th research visit, 7 days after last tDCS session and 8th visit 14 days after last tDCS session
  A visual search task will be given in which the participant looks for a T among L's. The contextual cuing task will consist of a practice block and forty test blocks. Eight of the trials in a block will consist of search configurations that repeat from block to block (repeat configurations); the other eight trials in a block will be randomly-generated configurations (new configurations). After the final trial, a recognition task will be presented to determine whether participants realized that repeat configurations were presented (not expected; cueing effects appear to result from implicit learning). Reaction time for each block will be recorded, with cognitive fatigue measured as deterioration of RT over the 40 blocks. This measure of change in RT will be compared across the 4 visits (pre-test, 6th visit, 7th visit, and 8th visit). Improved cognition fatigue based on tDCS treatment would predict reduced change in RT in the later visits compared to the pre-test.

SECONDARY OUTCOMES:
Change in Error Rate on contextual cueing computer task | 90 minutes; pre-test during the second research visit, post-test on 6th research visit after 5 consecutive days of tDCS, a follow up test on the 7th research visit, 7 days after last tDCS session and 8th visit 14 days after last tDCS session
  A visual search task will be given in which the participant looks for a T among L's. The contextual cuing task will consist of a practice block and forty test blocks. Eight of the trials in a block will consist of search configurations that repeat from block to block (repeat configurations); the other eight trials in a block will be randomly-generated configurations (new configurations). After the final trial, a recognition task will be presented to determine whether participants realized that repeat configurations were presented (not expected; cueing effects appear to result from implicit learning). Error rate for each block will be recorded, with cognitive fatigue measured as increased errors over the 40 blocks. This measure of change in error rate will be compared across the 4 visits (pre-test, 6th visit, 7th visit, and 8th visit). Improved cognition fatigue based on tDCS treatment would predict reduced change in error rate in the later visits compared to the pre-test.
Multidimensional Fatigue Inventory (MFI) | 5 minutes; pre-test during the second research visit, post-test on 6th research visit after 5 consecutive days of tDCS, a follow up test on the 7th research visit, 7 days after last tDCS session and 8th visit 14 days after last tDCS session
  This is a 20-item self-report instrument that measures five dimensions of fatigue independently: general fatigue, physical fatigue, mental fatigue, reduced motivation, and reduced activity.
Center for Epidemiological Studies Depression Scale (CES-D) | 5 minutes; pre-test during the second research visit, post-test on 6th research visit after 5 consecutive days of tDCS, a follow up test on the 7th research visit, 7 days after last tDCS session and 8th visit 14 days after last tDCS session
  This is a tool used to screen for symptoms of depression.
McGill Quality of Life (QOL) Scale | 1 minute; pre-test during the second research visit, post-test on 6th research visit after 5 consecutive days of tDCS, a follow up test on the 7th research visit, 7 days after last tDCS session and 8th visit 14 days after last tDCS session
  This is a single item tool to assess quality of life on all parts of life (physical, emotional, social, spiritual, and financial.
Neuropsychological battery (Stroop and Digit Span) | 10 minutes; pre-test during the second research visit, post-test on 6th research visit after 5 consecutive days of tDCS, a follow up test on the 7th research visit, 7 days after last tDCS session and 8th visit 14 days after last tDCS session
  The Stroop Test is a measure of processing speed, attention, and inhibition. In Stroop A, the participant is required to read color words (e.g., Red, Green, etc.) out loud quickly for 45 seconds. In Stroop B, the participant is required to name ink colors out loud as quickly as possible for 45 seconds. In Stroop C, the participants are required to name the color ink of opposing color words (e.g., the word "blue" written in red ink with the correct response being "red"). Digit Span forward is a measure of simple attention. Participants repeat progressively longer series of numbers until the participant can no longer complete the task. Digit Span Backward is a measure of working memory. The participant repeats back a series of numbers in reverse order. The series length increase until the participant can no longer complete the task.
Montreal Cognitive Assessment (MOCA) | 8 minutes; pre-test during the second research visit and post-test on 8th visit 14 days after last tDCS session
  This is a tool used to screen for mild cognitive dysfunctions. It assesses different domains of cognition: attention, memory, language visuospatial skills, orientation, and calculations.

CONTACTS AND LOCATIONS:
Overall Officials: Jau-Shin Lou, MD, Principal Investigator — Sanford Health
Locations (1):
- Sanford Brain & Spine Center, Fargo, North Dakota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Boggio PS, Ferrucci R, Rigonatti SP, Covre P, Nitsche M, Pascual-Leone A, Fregni F. Effects of transcranial direct current stimulation on working memory in patients with Parkinson's disease. J Neurol Sci. 2006 Nov 1;249(1):31-8. doi: 10.1016/j.jns.2006.05.062. Epub 2006 Jul 14. PMID 16843494
- [Background] Brunoni AR, Nitsche MA, Bolognini N, Bikson M, Wagner T, Merabet L, Edwards DJ, Valero-Cabre A, Rotenberg A, Pascual-Leone A, Ferrucci R, Priori A, Boggio PS, Fregni F. Clinical research with transcranial direct current stimulation (tDCS): challenges and future directions. Brain Stimul. 2012 Jul;5(3):175-195. doi: 10.1016/j.brs.2011.03.002. Epub 2011 Apr 1. PMID 22037126
- [Background] Lou JS, Kearns G, Oken B, Sexton G, Nutt J. Exacerbated physical fatigue and mental fatigue in Parkinson's disease. Mov Disord. 2001 Mar;16(2):190-6. doi: 10.1002/mds.1042. PMID 11295769
- [Background] Meinzer M, Jahnigen S, Copland DA, Darkow R, Grittner U, Avirame K, Rodriguez AD, Lindenberg R, Floel A. Transcranial direct current stimulation over multiple days improves learning and maintenance of a novel vocabulary. Cortex. 2014 Jan;50:137-47. doi: 10.1016/j.cortex.2013.07.013. Epub 2013 Aug 6. PMID 23988131
- [Background] Nitsche MA, Paulus W. Excitability changes induced in the human motor cortex by weak transcranial direct current stimulation. J Physiol. 2000 Sep 15;527 Pt 3(Pt 3):633-9. doi: 10.1111/j.1469-7793.2000.t01-1-00633.x. PMID 10990547